CLINICAL TRIAL: NCT04130035
Title: Decision Making in Degenerative Lumbar Spine: CT vs. MRI
Brief Title: Decision Making in Degenerative Lumbar Spine : CT vs. MRI
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Aamer, resident doctor, Assiut University
Other Study IDs: degenerative lumbar spine
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2019-10-17 (Actual); Status verified 2019-10

CONDITIONS: Degenerative Lumbar Disease
Keywords: decision making; degenerative lumbar disease; CT; MRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To identify the optimal imaging modality involved in decision making in patients with degenerative lumbar spine using CT vs. MRI.

DETAILED DESCRIPTION:
* There is 266 million individuals (3.63%) worldwide have DSD and LBP each year; the highest and lowest estimated incidences were found in Europe (5.7%) and Africa (2.4%), respectively. Based on population sizes, low- and middle-income countries have 4 times as many cases as high-income countries. Thirty-nine million individuals (0.53%) worldwide were found to have Spondylolisthesis, 403 million (5.5%) individuals worldwide with symptomatic disc degeneration, and 103 million (1.41%) individuals worldwide with spinal stenosis annually.
* Degenerative disease of the lumbar spine is a significant cause of disability in the world; it encompasses conditions such as Spondylolisthesis, disc degeneration, and lumbar spinal stenosis. Associated with a variety of clinical symptoms, including lower extremity pain, weakness, and low back pain (LBP) of varying levels of severity.
* Imaging plays an important role in the evaluation of degenerative spine.
* Plain films still play an important role in evaluation of the spine, because the examination is inexpensive and available and gives a wide panoramic view of the spine. Direct information about bony structures can be obtained, and functional information about misalignment and vertebral stability can be obtained with upright dynamic films in flexion-extension and lateral bending.
* Computerized axial tomography (CAT) scan: CT scan shows soft tissues such as ligaments and muscles more clearly than traditional X-rays do, so it is more useful for diagnosing certain problems, such as ruptured or degenerated discs and spinal stenosis.
* Magnetic resonance imaging (MRI): The advantage of MRI scans over X-rays and CT scans is that MRI provides clear, detailed images of the soft-tissue structures, such as the muscles, cartilage, ligaments, discs, tendons and blood vessels, in addition to the bones.

ELIGIBILITY:
Inclusion Criteria:

* degenerative lumbar spine diseases.
* age more than 18.

Exclusion Criteria:

* Patients with contraindications for MRI.
* Patients with spinal implants in the target region.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients more than 18 years old have degenerative lumbar disease with contraindication of MRI and have spinal implant at lumbar region.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2019-11-01 (Estimated); Primary Completion 2021-11-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
comparison between CT vs. MRI in decision making in degenerative lumbar spine. | baseline
  Differences in decision making in patients of lumbar degenerative spine based on CT vs. MRI.

SECONDARY OUTCOMES:
The correlation between the image finding and intraoperative finding. | baseline
  The correlation between the image finding and intraoperative finding.

CONTACTS AND LOCATIONS:
Overall Officials: essam Elsherief, prof., Study Chair — Assiut University

REFERENCES:
- [Background] Maravilla KR, Lesh P, Weinreb JC, Selby DK, Mooney V. Magnetic resonance imaging of the lumbar spine with CT correlation. AJNR Am J Neuroradiol. 1985 Mar-Apr;6(2):237-45. PMID 3920882
- [Background] Modic MT, Ross JS. Magnetic resonance imaging in the evaluation of low back pain. Orthop Clin North Am. 1991 Apr;22(2):283-301. PMID 1826552
- [Background] Jarvik JG, Deyo RA. Diagnostic evaluation of low back pain with emphasis on imaging. Ann Intern Med. 2002 Oct 1;137(7):586-97. doi: 10.7326/0003-4819-137-7-200210010-00010. PMID 12353946
- [Background] Ravindra VM, Senglaub SS, Rattani A, Dewan MC, Hartl R, Bisson E, Park KB, Shrime MG. Degenerative Lumbar Spine Disease: Estimating Global Incidence and Worldwide Volume. Global Spine J. 2018 Dec;8(8):784-794. doi: 10.1177/2192568218770769. Epub 2018 Apr 24. PMID 30560029